CLINICAL TRIAL: NCT03537365
Title: Bovine Colostrum to Fortify Human Milk for Preterm Infants A Randomized, Controlled Pilot Trial
Brief Title: Bovine Colostrum as a Fortifier Added to Human Milk for Preterm Infants
Acronym: FortiColos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Per Torp Sangild (Other)
Collaborators: Kolding Sygehus (Other); Herlev Hospital (Other); Hvidovre University Hospital (Other); Aarhus University Hospital (Other); Odense University Hospital (Other); Nordsjaellands Hospital (Other)
Responsible Party: Sponsor-Investigator, Per Torp Sangild, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FortiColos (pilot RCT)
Record Dates: First submitted 2018-01-16; First posted 2018-05-25 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Growth; Necrotizing Enterocolitis; Late-Onset Sepsis; Feeding Intolerance
Keywords: Human Milk Fortification; Bovine Colostrum; Very Preterm Infants; Enteral feeding; Human Milk; Neonatology; Colostrum
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A multicentre, non-blinded, pilot randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bovine Colostrum / intervention group (Experimental): Preterm infants are supplemented with bovine colostrum (BC) as a fortifier to human milk. BC is the first milk from cows after parturition and is a rich source of protein (80-150 g/L) and bioactive components, including lactoferrin, lysozyme, lactoperoxidase, immunoglobulins, and growth factors. The product is supplied in a sterile, powdered form and consists of unmodified, intact BC.
  Interventions: Dietary Supplement: Bovine Colostrum (BC) / intervention group
- FM85 / control group (Active Comparator): Preterm infants are supplemented with PreNAN FM85 as fortifier to human milk. PreNAN FM85 contains partially hydrolyzed protein and maltodextrin including vitamins and minerals. The product is supplied in a powdered form.
  Interventions: Dietary Supplement: FM85 / control group

INTERVENTIONS:
Dietary Supplement: Bovine Colostrum (BC) / intervention group — Infants randomized to the intervention group will receive a maximum of 2.8 g bovine colostrum (BC, Biofiber, Gesten, Denmark), as the HMF added to 100 ml of MM and/or DM, when EN has reached a dose of 100-140 ml/kg/d and blood urea nitrogen (BUN) levels are below 5 mmol/l.
  The infants starts with 1 g (0.5 g protein) BC per 100 ml human milk on the first day, increased to 2 g (1.0 g protein) on day 3, and finally 2.8 g (1.4 g protein) on day 5, if the infants only receive DM.
  The intervention begins if the infants meet the inclusions criteria and the intervention lasts until the infants reach post menstrual age (PMA) 34+6 weeks or are discharged home (including participating in an "early discharge program"), or are transferred to non-participating neonatal units, whichever comes first.
  Arms: Bovine Colostrum / intervention group
Dietary Supplement: FM85 / control group — Infants randomized to the control group will receive a maximum of 4 g PreNAN FM85 (Nestlé, Vevey, Switzerland) as HMF, added to 100 ml MM and/or DM, when EN has reached a dose of 100-140 ml/kg/d and BUN levels are below 5 mmol/l.
  The infants starts with 1 g (0.35 g protein) FM85 per 100 ml human milk on the first day, which will be increased to 3 g (1.05 g protein) on day 3 and finally 4 g (1.4 g protein) on day 5, if the infants only receive DM.
  FM85 is the standard HMF used in all participating hospitals in Denmark. The infants will receive FM85 as the HMF as long as additional protein in the milk is needed.
  Arms: FM85 / control group

SUMMARY:
Very preterm infants (<32 weeks gestation) with very low birth weight (VLBW, <1500 g) show immaturity of organs and have high nutrient requirements forgrowth and development. In the first weeks, they have difficulties tolerating enteral nutrition (EN) and are often given supplemental parenteral nutrition (PN). A fast transition to full EN is important to improve gut maturation and reduce the high risk of late-onset sepsis (LOS), related to their immature immunity in gut and blood. Conversely, too fast increase of EN predisposes to feeding intolerance and necrotizing enterocolitis (NEC). Further, human milk feeding is not sufficient to support nutrient requirements for growth of VLBW infants. Thus, it remains a difficult task to optimize EN transition, achieve adequate nutrient intake and growth, and minimize NEC and LOS in the postnatal period of VLBW infants.

Mother´s own milk (MM) is considered the best source of EN for VLBW infants and pasteurized human donor milk (DM) is the second choice, if MM is absent or not sufficient. The recommended protein intake is 4-4.5 g/kg/d for VLBW infants, when the target is a postnatal growth similar to intrauterine growth rates. This amount of protein cannot be met by feeding only MM or DM. Thus, it is common practice to enrich human milk with human milk fortifiers (HMFs, based on ingredients used in infant formulas) to increase growth, bone mineralization and neurodevelopment, starting from 7-14 d after birth and 80-160 ml/kg feeding volume per day. Bovine colostrum (BC) is the first milk from cows after parturition and is rich in protein (80-150 g/L) and bioactive components. These components may improve gut maturation, NEC protection and nutrient assimilation, even across species. Studies in preterm pigs show that feeding BC alone, or DM fortified with BC, improves growth, gut maturation and NEC resistance during the first 1-2 weeks, relative to DM, or DM fortified with conventional HMFs.On this background, we hypothesize that BC, used as a fortifier for MM or DM, can induce similar growth and better NEC and LOS resistance, than conventional fortifiers. A pilot trial is required 1) to test the feasibility and initial safety of BC as a fortifier (e.g. similar growth rates and clinical variables as conventional fortification), 2) to calculate the sample size for a later, larger RCT with NEC +LOS as the primary outcome, and 3) record paraclinical outcomes associated with type of fortifier.

DETAILED DESCRIPTION:
The main objectives of this multicentre, non-blinded, pilot, RCT are:

1. To investigate the safety, tolerability and the preliminary effects of BC, used as an HMF for MM and DM in very preterm infants.
2. To facilitate the determination of sample size for a later, larger RCT with NEC- and LOS-free survival as the primary outcome.
3. To assess the feasibility of study procedures, incl. recruitment rates, parental consent, adherence, sample collection, and clinical routines.

Participants Parents to eligible very preterm infants admitted to the Neonatal Intensive Care Units (NICU) at Nanshan People's Hospital (NAN) and Baoan Maternal and Children's Hospital in Shenzen, China will be asked for participation.

Since this is a pilot trial, a conventional sample size calculation, using only one primary outcome, is not required. The aim is to include 200 infants (100 per group), which is expected to give sufficient strength to demonstrate effects on the chosen feasibility outcomes and secondary blood and stool variables (see protocol). Statistical analyses will be performed blindly on both intention-to-treat and per protocol basis. Continuous outcomes will be summarized as mean and standard deviation (e.g., body weight) or median and interquartile range (e.g. time to reach full enteral feeding). Binary outcomes (e.g. incidence of NEC) will be presented as counts and percentages. To test the preliminary effects of BC, clinical and para-clinical outcomes will be compared between the two groups. The estimates will be presented as relative risk and absolute risk difference, difference between means, or hazard ratio, depending on the type of outcome. The estimates will be presented with a 95% confidence interval. Further statistical analyses are described in the protocol.

ELIGIBILITY:
Inclusion criteria:

1. Very preterm infants born between GA 26+0 and 30+6 weeks (from the first day of the mother's last menstrual period and/or based on fetal ultrasound)
2. DM is given at the unit when MM is absent (or insufficient in amount)
3. Infants judged by the attending physician to be in need of nutrient fortification, as added in the form of HMF to MM and/or DM
4. Infants admitted and staying at participating units at least until post menstrual age (PMA, gestational age + weeks and/or days since birth) 34+6 weeks, before being transferred to non-participating units, or going home participating in an "early discharge program". The infants can be transferred from one participating unit to another participating unit.

Exclusion criteria:

1. Major congenital anomalies and birth defects
2. Infants who have had gastrointestinal surgery prior to randomization
3. Infants who have received infant formula prior to randomization

Ages: 5 Days to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Body weight | From start of intervention to hospital discharge, or up to 14 weeks
  Weight gain in grams from birth to discharge from hospital. Weight at different time points will be calculated into z-scores according to a reference. Delta z-scores will be used to evaluate growth and for comparison between groups.
Incidence of necrotizing entercolitis (NEC) | From start of intervention to hospital discharge, or up to 14 weeks
  Number of infants in each group diagnosed with necrotizing enterocolitis (NEC) defined as Bell's stage II or above (Kliegman & Walsh 1987).
Incidence of late-onset sepsis (LOS) | From start of intervention to hospital discharge, or up to 14 weeks
  Number of infants in each group diagnosed with late-onset sepsis defined as clinical signs of infection >2 days after birth with antibiotic treatment for ≥5 days (or shorter than 5 days if the participant died) with or without one positive bacterial culture in blood or cerebral spinal fluid (CSF).

SECONDARY OUTCOMES:
Feeding intolerence | From start of intervention to end of study period at post menstrual age 34+6 weeks, or up to 8 weeks
  Proportion of days with a feeding volume less than 50% of the total planned volume per day
Time to reach full enteral feeding | From birth to full enteral feeding, or up to 8 weeks
  Number of days to full enteral feeding is reached - defined as the time when >150 ml/kg/d is reached and parenteral nutrition has been discontinued
Days on parenteral nutrition | From birth to end of intervention, or up to 8 weeks
  Number of days that the infant receives intravenous intakes of protein and/or lipid and/or glucose.
Length of hospital stay | From birth until until final discharge, or up to 14 weeks
  Number of days in hospital, defined as days from birth until final discharge (including the days covered by an early discharge programme).
Blood urea nitrogen (BUN) | Weekly from just before to end of intervention at postmenstrual age 34+6 weeks, or up to 8 weeks
  Blood urea nitrogen concentration is measured to evaluate the risk of excessive protein supply and immature kidney function
Blood minerals | Weekly from just before to end of intervention at postmenstrual age 34+6 weeks, or up to 8 weeks
  Blood levels of ionized phosphate, calcium and zink are measured to evaluate the risk of inadequate or excessive dietary mineral supply
Blood haemoglobin | Weekly from just before to end of intervention at postmenstrual age 34+6 weeks, or up to 8 weeks
  Determined to evaluate risk of anaemia and inadequate iron supply

OTHER OUTCOMES:
Body length | Weekly from just before to end of intervention at postmenstrual age 34+6 weeks, or up to 8 weeks
  Recorded as a measure of growth in cm by standardized measuring procedures
Head circumference | Weekly from just before to end of intervention at postmenstrual age 34+6 weeks, or up to 8 weeks
  Recorded as a measure of head growth in cm by standardized measuring procedures
Plasma amino acid levels | Prior to and after 1 and 2 weeks of intervention
  To determine whether individual amino acids are within their normal range. Specific attention is given to amino acids used as markers for excessive protein supply (tyrosine) and gut function (citrulline, arginine)
Plasma intestinal fatty acid binding protein (i-FABP) | Prior to and after 1 and 2 weeks of intervention
  Determine the concentration, as a marker of gut epithelial integrity
Plasma neutrophil extracellular trap (NET) components | Prior to and after 1 and 2 weeks of intervention
  Determine the concentration, as a marker systemic inflammation
Plasma lactoferrin | Prior to and after 1 and 2 weeks of intervention
  Determine the concentration, as a marker systemic inflammation
Plasma interleukin (IL) 8 | Prior to and after 1 and 2 weeks of intervention
  Determine the concentration, as a marker systemic inflammation
Fecal microbiota | Prior to and after 1 and 2 weeks of intervention
  Determine the 16S microbiome density and diversity, as a marker for gut microbiota stability
Fecal interleukin (IL) 8 | Prior to and after 1 and 2 weeks of intervention
  Determine concentration per g feces, as marker of gut inflammation
Fecal calprotectin (S100-A8/9) | Prior to and after 1 and 2 weeks of intervention
  Determine concentration per g faeces, as marker of gut inflammation
Fecal metabolites (short-chain fatty acids, SCFAs) | Prior to and after 1 and 2 weeks of intervention
  Determine concentration per g faeces, including acetate, butyrate and propionate levels, as markers of bacterial nutrient fermentation
Feasibility of study design | From study initiation to study completion at each participating hospital, data collected from each unit by the end of the study
  Record parental consent rates, infant recruitment rates, proportion of incomplete datasets
Feasibility of diet intervention | From study initiation to study completion at each participating hospital, data collected from each unit by the end of the study
  Determine by semi-quantitative questionaire evaluation, if the investigated BC product, relative to the control product, increases/decreases the work load or complications experienced by the involved clinical staff (doctors, nurses)

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Zachariassen, MD., PhD, Principal Investigator — Odense University Hospital; Per Sangild, Prof, Study Chair — Rigshospitalet, Denmark
Locations (7):
- Denmark (7):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet (RH), Copenhagen
  - Herlev Hospital, Herlev
  - North Zealand Hospital, Hillerød
  - Hvidovre Hospital (HH), Hvidovre
  - Kolding Hospital, Kolding
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang L, Hui Y, Sangild PT, Kot WP, Aunsholt L, Zachariassen G, Jiang P-P, Nielsen DS. Gut microbiota development in very preterm infants following fortification of human milk. mSystems. 2025 Mar 18;10(3):e0091624. doi: 10.1128/msystems.00916-24. Epub 2025 Feb 21. PMID 39982063
- [Derived] Lewis AE, Kappel SS, Hussain S, Sangild PT, Zachariassen G, Aunsholt L. Trial-related blood sampling and red blood cell transfusions in preterm infants. Acta Paediatr. 2023 Dec;112(12):2486-2492. doi: 10.1111/apa.16948. Epub 2023 Aug 16. PMID 37565393
- [Derived] Ahnfeldt AM, Hyldig N, Li Y, Kappel SS, Aunsholdt L, Sangild PT, Zachariassen G. FortiColos - a multicentre study using bovine colostrum as a fortifier to human milk in very preterm infants: study protocol for a randomised controlled pilot trial. Trials. 2019 May 22;20(1):279. doi: 10.1186/s13063-019-3367-7. PMID 31118098